CLINICAL TRIAL: NCT02983591
Title: Effect of Misoprostol in Reducing Post Partum Hemorrhage After Labor Induction by Oxytocin: a Prospective Randomized Controlled Trial
Brief Title: Effect of Misoprostol in Reducing Post Partum Hemorrhage After Labor Induction by Oxytocin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Manal Hubeish, OBGYN attending physician, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16082016
Record Dates: First submitted 2016-11-30; First posted 2016-12-06 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Prevention of Post Partum Hemorrhage After Labor Induction

ARMS (2):
- Misoprostol (Experimental): Rectal misoprostol
  Interventions: Drug: Misoprostol after delivery; Drug: Oxytocin before delivery
- Oxytocin (Experimental): intravenous oxytocin
  Interventions: Drug: Oxytocin after delivery; Drug: Oxytocin before delivery

INTERVENTIONS:
Drug: Misoprostol after delivery — Patients will receive 1000 mcg Misoprostol per rectum
  Arms: Misoprostol
Drug: Oxytocin after delivery — Patients will receive 20 units oxytocin intravenously in one liter of Lactated Ringer solution at a rate of 150ml/h
  Arms: Oxytocin
Drug: Oxytocin before delivery — All patients will receive oxytocin 0.5-1 milliUnit/min IV, titrated to 1-2 milliUnit/min every 15-60 min before delivery to induce labor

SUMMARY:
The use of Oxytocin for labor induction may cause receptor exhaustion and thus making its use in the third stage of labor ineffective in reducing post partum blood loss as compared to other uterotonics.So, we studied the effect of other uterotonic which is misoprostol in reducing post partum hemorrhage.

DETAILED DESCRIPTION:
Our study will be carried out at Makassed General Hospital, a tertiary-level maternity unit performing about 1000 deliveries annually. After approval by the hospital Ethics and Research Committee, women with single viable pregnancy, in cephalic presentation, at full term and whom labor was induced by Oxytocin will be eligible for inclusion.

After informed consents is obtained, the parturients will be assigned randomly according to a computer generated sequence in block lists of 25each time to receive either 1000mcg of Misoprostol rectally or 20 units of Oxytocin intravenously to run at a rate of 150ml/hr. The medications will be given just after cord clamping and before delivery of the placenta. Active management of the third stage of labor will be carried out simultaneously with early cord clamping, gentle downward traction of the placenta to hasten its delivery, and uterine massage in addition to the uterotonic according to assignment of the patient. Assessment of the uterine condition will be done by the obstetrician or his assistant, together with visually estimating the amount of blood loss. Once uterine atony or estimated blood loss (EBL) of more than 500 ml is noticed, another uterotonics will be administered according to the condition and at the discretion of the obstetrician.

Failure to achieve adequate uterine contraction and to control post partum hemorrhage (PPH) by the routine uterine massage will urge the use of either different uterotonics or surgical intervention if necessary. Blood transfusion will be ordered for the cases whose visual estimation of blood loss is more than 1000ml or when the patient was hemodynamically unstable. In order to compare the effect of each medication alone on the amount of blood loss, we will then exclude those patients who received blood transfusion or additional uterotonics. A base line hemoglobin and hematocrit levels will be withdrawn on admission and another reading 12 hours postpartum.

ELIGIBILITY:
Inclusion Criteria:

* women with single viable pregnancy,
* cephalic presentation,
* at full term
* whom labor was induced by Oxytocin were eligible

Exclusion Criteria:

* delivery by cesarean section
* received other prophylactic uterotonics

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2016-11; Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Hemoglobin level | 12 to 24 hours post partum
  10% or more drop in hemoglobin

SECONDARY OUTCOMES:
mean hemoglobin drop | 12 to 24 hours post partum
  difference between pre and post partum hemoglobin levels
mean estimated blood loss | during the first hour post partum
  visual estimation of blood loss
drop in hemoglobin | 12 to 24 hours post partum
  2g/dl drop in hemoglobin
side effect of medication | upto 48 hours after delivery
  fever > 38°C, diarrhea, and shivering

CONTACTS AND LOCATIONS:
Locations (1):
- Makassed General Hospital, Beirut, Lebanon